CLINICAL TRIAL: NCT04502082
Title: An Open-Label, Dose Escalation, Multi-Center Phase I/II Research Trial to Assess the Safety of ET140203 T Cells and Determine the Recommended Phase II Dose (RP2D) in Adults With Advanced Hepatocellular Carcinoma (HCC) (ARYA-1)
Brief Title: Study of ET140203 T Cells in Adults With Advanced Hepatocellular Carcinoma (ARYA-1)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was intended to be a Phase 1/2 trial, but the sponsor terminated the trial prior to moving to Phase 2 to direct efforts to the pediatric study (ARYA-2) for this product.
Sponsor: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETUS19AFPAR121
Record Dates: First submitted 2020-07-22; First posted 2020-08-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasm; Metastatic Liver Cancer
Keywords: Hepatocellular Carcinoma HCC; Advanced HCC; Late-Stage HCC; Liver Cancer; Liver Neoplasm; Metastatic Liver Cancer; Metastatic HCC; T-cell therapy; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ET140203 TCells (Experimental): ET140203 T Cells
  Interventions: Biological: ET140203 autologous T cell product

INTERVENTIONS:
Biological: ET140203 autologous T cell product — Autologous T cells transduced with lentivirus encoding an ET140203 expression construct

SUMMARY:
Open-label, dose escalation, multi-center, Phase I / II study to assess the safety of an autologous T-cell product (ET140203) in adult subjects with Alpha-fetoprotein (AFP)-positive/Human Leukocyte Antigen (HLA) A-2-positive advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The purpose of this study is to investigate an autologous T-cell therapy for advanced hepatocellular carcinoma (HCC). ET140203 T cells are autologous T cells genetically modified to carry a TCR-mimic (TCRm) construct capable of mediating cell killing by targeting tumor specific intracellular antigens and addressing solid tumor therapy challenges.

The trial was intended to be a Phase 1/2 trial, but the sponsor terminated the trial prior to moving to Phase 2 to direct their efforts to the pediatric study (ARYA-2) for this product.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC with serum AFP >100ng/ml at time of screening and following most current line of therapy OR radiographic diagnosis of HCC with serum AFP >400ng/ml at time of screening and following most current line of therapy.
* Metastatic or locally advanced, unresectable HCC
* Must have failed or not tolerated at least two (2) different anti-HCC systemic agents
* Molecular Human Leukocyte Antigen ("HLA") class I allele typing confirms participant carries at least one HLA-A2 allele
* Life expectancy of at least 4 months
* Karnofsky Performance Scale greater than or equal to 70
* At least 1 measurable lesion on imaging by RECIST
* Child-Pugh A6 or better
* Absolute neutrophil count greater than or equal to 1,500/mm^3
* Platelet count greater than or equal to 75,000/mm^3

Exclusion Criteria:

* Clinically significant cardiac disease
* Clinically significant pre-existing illness or active infection
* Clinically significant Central Nervous System (CNS) or neural dysfunction
* Active autoimmune disease requiring therapy
* Active malignancy other than HCC with the exception of cholangiocarcinoma (CCA) or any malignancy with an expected survival ≥ 3 years without any treatment (exception: hormone/androgen-deprivation therapy) and without any organ involvement
* History of organ transplant
* Compromised circulation in portal vein, hepatic vein, or vena cava due to obstruction
* Advanced HCC involving greater than 50% of the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence rates of adverse events (AEs) after infusion of ET140203 T cells | 28 days
  Safety of ET140203T cells as assessed by the number of adverse events (AEs) after infusion
Severity rates of adverse events (AEs) after infusion of ET140203 T cells | 28 days
  Safety of ET140203T cells as assessed by the severity of adverse events (AEs) after infusion.
Incidence rates of dose limiting toxicities (DLTs) after infusion of ET140203 T cells | 28 days
  Tolerability of ET140203T cells after infusions assessed by committee review of dose limiting toxicities (DLTs)
The recommended phase 2 dose (RP2D) regimen of ET140203 T-cell therapy primarily based on DLT | up to 2 years
  The RP2D will be determined by the study Dose Escalation Committee (DEC) and primarily based on DLT, and secondarily on the best tumor response

SECONDARY OUTCOMES:
Assess the efficacy of ET140203 T cells in adults with advanced HCC. | up to 2 years
  Response rate will be assessed by radiographic scans and assessed according to RECIST criteria.
Determine the pharmacokinetics of ET140203 T cells after infusion. | up to 2 years
  Assess the persistence of ET140203 T cells circulating in blood over time

CONTACTS AND LOCATIONS:
Overall Officials: Pei Wang, PhD, Study Director — Eureka Therapeutics Inc.
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Kansas University Medical Center, Westwood, Kansas

IPD SHARING:
Plan to Share IPD: No